CLINICAL TRIAL: NCT01644045
Title: Prehospital Emergency Care of Obstructive Respiratory Emergencies With the Use of Teleconsultation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 005-1003-0034-4; PtJ-Az.: z0909im002b (Other Grant/Funding Number: PTJ)
Record Dates: First submitted 2012-07-12; First posted 2012-07-18 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-09

CONDITIONS: Asthma; COPD
Keywords: Asthma; COPD; emergency medical service; teleconsultation; telemedicine
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Device: Teleconsultation (Experimental): In cases of acute obstructive, respiratory emergencies if patients give informed consent the paramedics can use this system to contact a so called "tele-EMS physician" who has an audio-connection to the EMS team and receives vital parameters (e.g., ECG, pulse oximetry, non-invasive blood pressure) in real-time. The transmission of still pictures (taken with a smartphone), 12-lead-ECGs and video streaming from the inside of the ambulance can also be carried out, if indicated. The tele-EMS physician supports the EMS team in obtaining all relevant medical history, diagnosis and can delegate the application of medications. This can be carried out to bridge the time to the arrival of an EMS physician or in less severe cases without an EMS physician on-scene. The quality of prehospital care and the possible influences on the initial inhospital phase should be investigated and compared with regular EMS.
  Interventions: Device: Teleconsultation

INTERVENTIONS:
Device: Teleconsultation — Teleconsultation for the EMS in acute respiratory emergencies

SUMMARY:
The aim of the study is to investigate the quality of prehospital emergency care in acute respiratory emergencies, when paramedics are supported telemedically by an EMS physician.

DETAILED DESCRIPTION:
Six ambulances from five different Emergency Medical Service (EMS) districts are equipped with a portable telemedicine system. In cases of acute obstructive, respiratory emergencies the paramedics can use this system to contact a so called "tele-EMS physician" after consent of the patient was obtained. The tele-EMS physician has an audio-connection to the EMS team and receives vital parameters (e.g., ECG, pulse oximetry, non-invasive blood pressure) in real-time. The transmission of still pictures (taken with a smartphone), 12-lead-ECGs and video streaming from the inside of the ambulance can also be carried out, if indicated. The tele-EMS physician supports the EMS team in obtaining all relevant medical history, diagnosis and can delegate the application of medications. This can be carried out to bridge the time to the arrival of an EMS physician or in less severe cases without an EMS physician on-scene. The quality of prehospital care and the possible influences on the initial inhospital phase should be investigated and compared with regular EMS.

ELIGIBILITY:
Inclusion Criteria:

* Obstructive, respiratory emergency
* Verbal consent for teleconsultation obtained or patient is not able to consent due the severity of the emergency

Exclusion Criteria:

* No respiratory emergency
* Refused consent for teleconsultation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-08; Primary Completion 2013-07 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Oxygen Saturation | average 1 hour
  Measurement of pulse oximetric oxygen saturation at the timepoint of first contact with a physician (EMS physician OR hospital arrival)

SECONDARY OUTCOMES:
Quality of emergency care | average 1 hour
  Analysis of the quality of prehospital care on the basis of published guidelines for asthma / COPD.
Rate of ventilation | average 1 hour
  Fraction of patients that receive invasive or non-invasive ventilation during the prehospital phase
Rate of complications | 2 hours
  Rate of complications due to medications: allergic reaction, heart rhythm problems

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Rossaint, Prof. Dr., Study Chair — University Hospital Aachen, Germany, Department of Anesthesiology; Jörg C Brokmann, Dr., Principal Investigator — University Hospital Aachen, Germany, Emergency Department
Locations (1):
- University Hospital Aachen, Aachen, Germany